CLINICAL TRIAL: NCT01526226
Title: Patient Comfort During High Flow Nasal Cannula (HFNC)Versus Nasal Continuous Airway Pressure (CPAP): a Cross Over Randomised Trial
Brief Title: Patient Comfort During High Flow Nasal Cannula Versus Nasal Continuous Airway Pressure (CPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-2019 REK NORD
Record Dates: First submitted 2012-01-02; First posted 2012-02-03 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2013-06

CONDITIONS: Respiratory Distress Syndrome, Newborn; Medical Device Discomfort
Keywords: High flow nasal cannula; Discomfort
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFNC (Experimental): High flow nasal cannula
  Interventions: Device: Respiratory support HFNC; Device: Respiratory support NCPAP
- nCPAP (Active Comparator): Nasal CPAP
  Interventions: Device: Respiratory support HFNC; Device: Respiratory support NCPAP

INTERVENTIONS:
Device: Respiratory support HFNC — In the cross over study 2 types of respiratory support are compared; HFNC versus nCPAP
  Other Names: HFNC; Fisher and Paykel
Device: Respiratory support NCPAP — In the cross over study 2 types of respiratory support are compared; HFNC versus nCPAP
  Other Names: NCPAP: Infant Flow (CareFusion)

SUMMARY:
Preterm children are at increased risk for developing lung disease due to immature lungs. Non-invasive ventilation (NIV) support is increasingly used as treatment. Nasal continuous positive airway pressure (nCPAP) is the most common NIV-mode. Recently, high flow nasal cannulas (HFNC) have become an alternative NIV-mode. Both nCPAP and HFNC provide increased pressure in the airways aiming to keep the lungs open. With nCPAP it is common to use short binasal prongs that fill the nostrils completely and are pressed tightly over the nose. With HFNC oxygen/air is administered via two small, thin cannulas located just inside the nostrils, but the nostrils are not blocked.

The aim of this study is to compare patient comfort in premature infants treated with nCPAP and HFNC. The investigators hypothesis is that HFNC increases patient comfort.

The study is a randomized cross over study (2 x 24 hours). Children eligible for inclusion should be born before 34 weeks of gestation and have moderate respiratory distress, thus be "in need" of nCPAP. During the study period (48 hours) the investigators will consider how the child tolerates treatment with nCPAP versus HFNC. Primary outcome is patient comfort assessed with the EDIN-score (Neonatal pain and comfort score). Secondary outcomes are stress hormone response (cortisol in saliva), surrounding noise and parental satisfaction. The child's breathing pattern will be carefully monitored. The study involves no extra painful investigations.

The investigators plan to recruit 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to the NICU at University Hospital of North Norway, Tromsoe, Norway (single center study)

  * Gestational age (GA) < 34 weeks
  * Corrected age < 34 weeks
  * Receiving nasal CPAP for respiratory distress
  * Respiratory "stable": FiO2 < 30%, pCO2 < 8,5 kPa and pH > 7.25.
* GA < 29 weeks: Respiratory "stable" over last 72 h.
* GA 29-33 weeks: Respiratory "stable" over last 24 h.

Exclusion Criteria:

1. Congenital anomalies
2. Ongoing treatment for hypoglycemia or infection
3. Other intercurrent disease requiring frequent blood sampling

Ages: 25 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Patient comfort (EDIN score) | 48 h (CPAP 24 h and HFNC 24 h); cumulative EDIN score for each 24 epoch is calculated and a change between the two interventions are assessed
  EDIN score (neonatal pain and comfort score) is a validated scoring system to assess pain and comfort in term and preterm infants. The cumulative EDIN score, based on three evaluations/24 h, is recorded for each 24 h epoch with HFNC or CPAP, respectively. The change in EDIN score between the two 24 h epochs are assessed.

SECONDARY OUTCOMES:
Noise | Measured at 10 AM and 10 PM over 48 h (4 measurements)
  Surrounding noise (dB)is measured twice daily during the 2 x 24 (48) h study period; twice during CPAP and twice during HFNC.
Parental satisfaction | Three questions answered after 24 h and 48 h
  3 questions related to parental satisfaction are asked by the end of each 24 h epoch with either CPAP or HFNC.
Stress hormone response (salivary cortisol) | Measured at 10 AM and 10 PM over 48 h (4 measurements)
  Salivary cortisol is used as a marker of stress hormone response. Salivary cortisol is collected twice (10 AM and 10 PM) for every 24 h epoch; a total of 4 measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Klingenberg, MD, PhD, Principal Investigator — University Hospital of North Norway, Tromsø, Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Background] Wilkinson D, Andersen C, O'Donnell CP, De Paoli AG. High flow nasal cannula for respiratory support in preterm infants. Cochrane Database Syst Rev. 2011 May 11;(5):CD006405. doi: 10.1002/14651858.CD006405.pub2. PMID 21563154
- [Derived] Klingenberg C, Pettersen M, Hansen EA, Gustavsen LJ, Dahl IA, Leknessund A, Kaaresen PI, Nordhov M. Patient comfort during treatment with heated humidified high flow nasal cannulae versus nasal continuous positive airway pressure: a randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F134-7. doi: 10.1136/archdischild-2013-304525. Epub 2013 Nov 13. PMID 24225220